CLINICAL TRIAL: NCT03709238
Title: Pain Processing and Pain Reporting in Patients With Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: UAarhus_Susan
Record Dates: First submitted 2018-09-03; First posted 2018-10-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-05

CONDITIONS: Pain
Keywords: Pain; Alzheimers disease
MeSH Terms: conditions — Pain; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimers diseased patients: Behavioral: Different thermal stimulation. Recording of facial expression during thermal stimulation.
  Interventions: Behavioral: Thermal stimulation
- Healthy participants: Behavioral: Different thermal stimulation. Recording of facial expression during thermal stimulation.
  Interventions: Behavioral: Thermal stimulation

INTERVENTIONS:
Behavioral: Thermal stimulation — Thermal stimulation

SUMMARY:
The study investigates pain processing and pain reporting in patients with Alzheimers disease compared to healthy participants.

Employing a within-subject design, the study includes patients with Alzheimers disease and healthy participants that are exposed to thermal stimuli. During the test session the facial expressions of the participant are video recorded.

By repeating this on separate test days, the involvement of pain relief and pain increase is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate patients with Alzheimers disease (group 1)
* Healthy participants ( group 2)

Exclusion Criteria:

* Chronic pain conditions
* Other medical, psychiatric or neurological disorders
* Use of pain-reliving medication 24 hours prior to testing

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with Alzheimers disease
  2. Healthy participants
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Participants will be tested on three different days. The numerical rating scale will be applied after each thermal stimulus for each test session.
  Acute pain assessed on numerical rating scale from 0 (no pain experience) to 10 (worst pain), examining pain intensity. The participant will provide a number on the scale which reflects their pain intensity.

SECONDARY OUTCOMES:
Pain Assessment in persons with Impaired Cognition (PAIC) | Participants will be video recorded on each of the three test days during testing.
  Video recordings will be analyzed with the PAIC scale from 0 (not at all) to 3 (great degree).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology and Behavioural Sciences, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matthiesen ST, Sieg M, Andersen SS, Amanzio M, Finnerup NB, Jensen TS, Gottrup H, Vase L. Placebo analgesia and nocebo hyperalgesia in patients with Alzheimer disease and healthy participants. Pain. 2024 Feb 1;165(2):440-449. doi: 10.1097/j.pain.0000000000003035. Epub 2023 Sep 8. PMID 37703397